CLINICAL TRIAL: NCT07256275
Title: Examining Peer Influences in Alcohol and Sexual Violence Among Marines Using a Dyadic Multimethod Approach
Brief Title: Peer Influences in Alcohol and Sexual Violence Among Marines Dyads
Status: Not yet recruiting | Type: Observational
Sponsor: Georgia State University (Other)
Collaborators: Medical University of South Carolina (Other); University of Colorado Health (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Amanda Gilmore, Associate Professor, Georgia State University
Other Study IDs: H25332
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Peer Influence; Alcohol-Involved Sexual Violence Perpetration
Keywords: Alcohol-Involved Sexual Violence Perpetration; Ecological Momentary Assessment; Sexual Imposition Task; Peer Influence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Confederate Group: Intoxicated Man: Participants in this group are randomly assigned to complete the experiment with a confederate who is an intoxicated man.
- Confederate Group: Sober Man: Participants in this group are randomly assigned to complete the experiment with a confederate who is a sober man.
- Confederate Group: Intoxicated Woman: Participants in this group are randomly assigned to complete the experiment with a confederate who is an intoxicated woman.
- Confederate Group: Sober Woman: Participants in this group are randomly assigned to complete the experiment with a confederate who is a sober woman.

SUMMARY:
The goal of this experimental study is to examine the complex and multifaceted influence of peers on alcohol-involved sexual violence perpetration (ASVP) in U.S. Marine Corps (USMC) men. The specific aims are:

Aim 1: Use ecological momentary assessment (EMA) to examine event-level effects of one's own alcohol use, peer alcohol use, and injunctive norms on ASVP intentions among dyads of Marine men who drink together (n=160 dyads; 320 total participants).

Aim 2: Examine the individual and peer effects on ASVP behavior in an experimental paradigm with a gender x confederate (potential victim) intoxication status design. In-the-moment dyad-peer verbalized encouragement for ASVP ("go cues") will be assessed by qualitatively coding verbalizations during the interaction.

Aim 3: Examine modifiable risk factors on ASVP intentions in vivo (Aim 1; EMA) and ASVP behavior in vitro (Aim 2; experiment) settings.

Participants will complete: 1) an individual orientation session with informed consent, baseline assessment, and EMA demo; 2) 14 days of EMA completed individually; and 3) a dyadic session to complete an experimental paradigm via videoconferencing. All study procedures will be completed in off-duty time as to not interfere with military duties.

DETAILED DESCRIPTION:
The overarching goal of this R01 is to obtain an event-level understanding of the role of alcohol and peer interpersonal behavior in sexual violence perpetration among Marine men. Rates of heavy episodic drinking and military sexual assault are high in the military, and highest among Marines. Alcohol is involved in 21-80% of sexual violence incidents among servicewomen and 14-56% of incidents among servicemen. Perceived peer norms and interpersonal interactions are key predictors of alcohol use and alcohol-involved sexual violence perpetration (ASVP) among civilians; however, it is unclear if these risk factors operate similarly in military populations. Peers in the US Marine Corps are unique and exert powerful influence on adaptive behaviors and attitudes and more negative health behaviors such as alcohol misuse. The proposed multi-method project, implemented by an experienced team of investigators, will simultaneously address several major and persistent gaps in knowledge. First, the investigators will obtain an event-level understanding of the effects of one's own and peer alcohol use, and the role of alcohol in ASVP norms on ASVP intentions in the US Marine Corps by integrating findings from in vivo and in vitro assessment methods. Second, this study will examine and assess the individual and peer effects of in-the-moment encouragement and discouragement on ASVP behaviors in an experimental paradigm. The investigators will accomplish this by leveraging innovative dyadic approaches employed among civilian dyads, thereby elucidating peer influences on ASVP among men in the US Marine Corps. The proposed study will recruit pairs of enlisted men currently serving in the US Marine Corps who engaged in heavy episodic drinking at least twice together in the past month. Dyads will complete ecological momentary assessments about their own and perceived peer alcohol use and ASVP intentions twice daily for 14 days. The study will also compare modifiable risk effects of peer influence acceptance of ASVP intentions and behaviors in vivo and in vitro settings.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged 21 or older
* Currently serving in the United States Marine Corps (USMC)
* Marine dyads must have engaged in heavy episodic drinking (≥5 drinks in less than two hours) together at least twice in the past month
* Marine dyads must rate their peer at a minimum of "somewhat important" on the Important People Interview.

Exclusion Criteria:

* The only exclusion criteria is not meeting inclusion criteria.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Study Population: Men aged 21 or older who drink alcohol and are currently serving in the United States Marine Corps (USMC).
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Sexual Strategies Survey | For 14 days after enrollment
  Alcohol-involved sexual violence intentions will be assessed using a modified version of the Sexual Strategies Survey. Scores range from 0-168, higher scores indicate higher intentions.
Sexual Experiences Survey-Long Form Perpetration - Noncontact Items | For 14 days after enrollment
  Alcohol-involved sexual violence intentions will be assessed using the noncontact items from the Sexual Experiences Survey-Long Form Perpetration (SES-LFP). Scores range from 0-49, higher scores indicate higher intentions.
Sexual Imposition Task | Experiment at 14 days after enrollment
  Alcohol-involved sexual violence perpetration behavior will be assessed using the Sexual Imposition Task. Choice of film and duration of clip will both be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K Gilmore, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data, only de-identified data.

DOCUMENTS (1):
  • Informed Consent Form (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT07256275/ICF_000.pdf